CLINICAL TRIAL: NCT02725593
Title: A 24 Week, Multicenter, Randomized, Double-Blind, Parallel Group, Phase 3 Trial With a 28 Week Long Term Safety Extension Period Evaluating the Safety and Efficacy of Dapagliflozin 10 mg in T2DM Patients Aged 10-24 Years
Brief Title: Study to Evaluate Safety and Efficacy of Dapagliflozin in Patients With Type 2 Diabetes Mellitus Aged 10-24 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry); Q2 Solutions (Industry); PRA Health Sciences (Industry); Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1690C00017; 2015-005041-31 (EudraCT Number)
Record Dates: First submitted 2016-03-29; First posted 2016-04-01 (Estimated); Results first posted 2020-12-02 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-01

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes Mellitus; Dapagliflozin; Placebo; Insulin resistance; Metabolic Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance; Metabolic Diseases | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dapagliflozin (Experimental)
  Interventions: Drug: Dapagliflozin
- Dapagliflozin placebo (Placebo Comparator)
  Interventions: Drug: Dapagliflozin placebo

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin 10 mg tablets administered orally once daily, for the 24-week blinded treatment period. Dapagliflozin 10mg tablets administered orally once daily, for the 28-week site and subject blinded long term extension.
  Other Names: FORXIGA
  Arms: Dapagliflozin
Drug: Dapagliflozin placebo — matching placebo tablets, administered orally once daily, for the 24-week blinded treatment period. Dapagliflozin 10mg tablets administered orally once daily,for the 28-week site and subject blinded long term extension.
  Arms: Dapagliflozin placebo

SUMMARY:
A trial of patients aged 10-24 years with type 2 diabetes mellitus to evaluate the comparative efficacy and safety between dapagliflozin and Placebo.

DETAILED DESCRIPTION:
A 24 Week, Multicenter, Randomized, Double-Blind, Parallel Group, Phase 3 Trial with a 28 Week Long Term Safety Extension Period Evaluating the Safety and Efficacy of Dapagliflozin 10 mg in T2DM Patients aged 10-24 years

ELIGIBILITY:
Inclusion Criteria

1. Provision of informed consent prior to any study-specific procedures
2. Males and Females, ages 10 years of age, up to but not including 25 years of age at the time of randomization
3. Previously diagnosed as having type 2 diabetes for at least 2 months by WHO/ADA diagnostic criteria
4. HbA1c >= 6.5% and <= 11% obtained at screening visit
5. Currently on diet and exercise and a stable dose of metformin (at least 1000 mg daily) for a minimum of 8 weeks, or stable dose of insulin for a minimum of 8 weeks, or a stable combination of metformin (at least 1000 mg daily) and insulin for a minimum of 8 weeks prior to screening
6. FPG <=255 mg/dL (<= 14.2 mmol/L) obtained at screening visit

Exclusion Criteria:

1. Previous diagnosis of Type 1 diabetes
2. Diabetes ketoacidosis (DKA) within 6 months of screening
3. Current use of the following medications for the treatment of diabetes, or use within the specified timeframe prior to screening for the main study:

   * Eight weeks: sulfonylureas, alpha glucosidase inhibitors, metiglinide, or injectable incretins or incretin mimetics or other antidiabetes medications not otherwise specified
   * Sixteen weeks: thiazolidinediones
   * Any previous history or current use of an SGLT2 inhibitor, including dapagliflozin
4. Initiation or discontinuation of prescription or non-prescription weight loss drugs within 8 weeks of screening.

   Use of prescription or non-prescription weight loss drugs must be stable during the study
5. Pregnant, positive serum pregnancy test, planning to become pregnant during the clinical trials, or breastfeeding
6. History of unstable or rapidly progressive renal disease
7. History of unresolved vesico-ureteral reflux
8. Replacement or chronic systemic corticosteroid therapy, defined as any dose of systemic corticosteroid taken for > 4 weeks within 3 months prior to the Day 1 visit.

   Note: Topical, nasal, or inhaled corticosteroids are allowed
9. Abnormal renal function, which is defined in subjects < 18 years of age as an estimated glomerular filtration rate (eGFR) calculated by the Schwartz Formula < 80 mL/min/1.73 m2 (1.33 mL/s), and in subjects >= 18 years as an estimated glomerular filtration rate (eGFR) calculated by the MDRD Formula < 60 mL/min/1.73 m2 (1.33 mL/s)
10. Presence of either: antibodies to glutamic acid decarboxylase (GAD) or protein tyrosine phosphatase-like protein antibodies (IA-2)
11. An abnormal TSH value at screening will be further evaluated for free T4. Subjects with abnormal free T4 values will be excluded
12. Hematuria (confirmed by microscopy at screening) with no explanation as judged by the investigator up to randomization
13. Anemia of any etiology defined as hemoglobin <=10.7 g/dL (107 g/L) for females and <= 11.3 g/dL (113 g/L) for males. Subjects who are considered to have anemia according to local guidelines should be excluded
14. Volume-depleted subjects. Subjects at risk for volume depletion due to co-existing conditions or concomitant medications, such as loop diuretics, should carefully monitor their volume status

Ages: 10 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-04-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (41):
- United States (14):
  - Research Site, New Haven, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Gainesville, Florida
  - Research Site, Homestead, Florida
  - Research Site, Miami, Florida
  - Research Site, Boston, Massachusetts
  - Research Site, Buffalo, New York
  - Research Site, The Bronx, New York
  - Research Site, Columbus, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Greenville, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Lampasas, Texas
  - Research Site, McAllen, Texas
- Hungary (2):
  - Research Site, Budapest
  - Research Site, Nyíregyháza
- Israel (5):
  - Research Site, Beersheba
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Ramat Gan
  - Research Site, Ẕerifin
- Mexico (6):
  - Research Site, Culiacán
  - Research Site, Guadalajara
  - Research Site, Mérida
  - Research Site, México, D.F.
  - Research Site, Monterrey
  - Research Site, Zapopan
- Romania (2):
  - Research Site, Oradea
  - Research Site, Timișoara
- Russia (10):
  - Research Site, Izhevsk
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Pyatigorsk
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Saratov
  - Research Site, Tomsk
- United Kingdom (2):
  - Research Site, Kent
  - Research Site, Leicester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Tamborlane WV, Laffel LM, Shehadeh N, Isganaitis E, Van Name M, Ratnayake J, Karlsson C, Norjavaara E. Efficacy and safety of dapagliflozin in children and young adults with type 2 diabetes: a prospective, multicentre, randomised, parallel group, phase 3 study. Lancet Diabetes Endocrinol. 2022 May;10(5):341-350. doi: 10.1016/S2213-8587(22)00052-3. Epub 2022 Apr 1. PMID 35378069
- See also: D1690C00017_CSP_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1690C00017&attachmentIdentifier=a9e77cda-496a-4e09-aa87-cbe0538b927b&fileName=D1690C00017_CSP_redacted.pdf&versionIdentifier=
- See also: D1690C00017_SAP_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1690C00017&attachmentIdentifier=27e64a31-b91e-45ea-bd34-12f4c16b9806&fileName=D1690C00017_SAP_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 42 study centres in 7 countries worldwide.
Groups:
- Dapagliflozin 10mg/ Dapagliflozin 10mg: Dapagliflozin (10 mg) tablet administered orally, once daily for the 24 week double-blinded treatment period. The participants then continued to receive Dapagliflozin (10 mg) once daily for a further 28 weeks in the open label long term-extension.
- Placebo/ Dapagliflozin 10mg: Matching placebo tablet administered orally, once daily for the 24 weeks double-blinded treatment period. The participants then received Dapagliflozin (10 mg), orally, once daily for a further 28 weeks in the open label long-term extension.
Period: Blinded Treatment Period
Arm/Group | Dapagliflozin 10mg/ Dapagliflozin 10mg | Placebo/ Dapagliflozin 10mg
Started | 39 | 33
Received Treatment | 39 | 33
Completed | 34 | 27
Not Completed | 5 | 6
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Withdrawal by Parent/Guardian | 0 | 2
Not completed — Lost to Follow-up | 1 | 1
Period: Long Term Extension
Arm/Group | Dapagliflozin 10mg/ Dapagliflozin 10mg | Placebo/ Dapagliflozin 10mg
Started | 33 (1 participant who completed Period 1 did not enter the long-term extension period.) | 27
Completed | 32 | 24
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin 10mg/ Dapagliflozin 10mg | Placebo/ Dapagliflozin 10mg | Total
Number analyzed (Participants) | 39 | 33 | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 16.1 (3.3) | 16.2 (3.6) | 16.1 (3.4)
Age, Customized [Count of Participants; unit: Participants]
  ≥10 and ≤15 | 16 | 14 | 30
  >15 and <18 | 13 | 10 | 23
  ≥18 and <25 | 10 | 9 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 19 | 43
  Male | 15 | 14 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 12 | 24
  Not Hispanic or Latino | 26 | 21 | 47
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 28 | 16 | 44
  Black or African American | 8 | 10 | 18
  Asian | 0 | 1 | 1
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  American Indian or Alaska Native | 2 | 3 | 5
  Other | 0 | 3 | 3
Geographic Region [Count of Participants; unit: Participants]
  North America | 16 | 16 | 32
  Latin America | 7 | 9 | 16
  Europe | 16 | 8 | 24
  Asia/Pacific | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Change From Baseline in Glycated Haemoglobin (HbA1c) at Week 24
Time Frame: Baseline to Week 24
Population: Full analysis set: All participants who were randomized and assigned to a treatment group, with baseline and at least one-post baseline value, prior to rescue therapy initiation or discontinuation from study treatment.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Dapagliflozin 10mg/ Dapagliflozin 10mg | Placebo/ Dapagliflozin 10mg
Number analyzed (Participants) | 31 | 23
Percentage of HbA1c | -0.25 (0.30) | 0.50 (0.34)
Statistical Analysis 1: Comparison: Dapagliflozin 10mg/ Dapagliflozin 10mg vs Placebo/ Dapagliflozin 10mg; Test type: Superiority; p = 0.101, Mixed model repeated measures analysis; Mean Difference (Final Values) = -0.75, 95% CI 2-sided [-1.65 to 0.15], Standard Error of Mean 0.45

2. Secondary Outcome: Adjusted Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Dapagliflozin 10mg/ Dapagliflozin 10mg | Placebo/ Dapagliflozin 10mg
Number analyzed (Participants) | 31 | 23
mmol/L | -0.07 (0.53) | 0.72 (0.61)
Statistical Analysis 1: Comparison: Dapagliflozin 10mg/ Dapagliflozin 10mg vs Placebo/ Dapagliflozin 10mg; Test type: Superiority; p = 0.340, Mixed model repeated measures analysis; Mean Difference (Final Values) = -0.78, 95% CI 2-sided [-2.42 to 0.85], Standard Error of Mean 0.81

3. Secondary Outcome: Percentage of Participants Who Required Glycemic Rescue Medication or Permanently Discontinued Treatment Due to Lack of Glycemic Control
Time Frame: Baseline to Week 24
Population: Full analysis set: All participants who were randomized and assigned to a treatment group.
Measure: Number; unit: Percentage of participants
Arm/Group | Dapagliflozin 10mg/ Dapagliflozin 10mg | Placebo/ Dapagliflozin 10mg
Number analyzed (Participants) | 39 | 33
Percentage of participants | 5.1 | 9.1
Statistical Analysis 1: Comparison: Dapagliflozin 10mg/ Dapagliflozin 10mg vs Placebo/ Dapagliflozin 10mg; Test type: Superiority; p = 0.655, Fisher's exact test; Mean Difference (Final Values) = -3.96, 95% CI 2-sided [-20.11 to 9.62]

4. Secondary Outcome: Percentage of Participants With Baseline Glycated Haemoglobin (HbA1c) >= 7% Who Achieved HbA1c Level < 7% at Week 24
Time Frame: Baseline to Week 24
Population: Full analysis set: All participants who were randomized and assigned to a treatment group, with HbA1c >=7% at baseline, with baseline and at least one-post baseline value, prior to rescue therapy initiation or discontinuation from study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Dapagliflozin 10mg/ Dapagliflozin 10mg | Placebo/ Dapagliflozin 10mg
Number analyzed (Participants) | 28 | 24
Percentage of participants | 25.0 | 4.2
Statistical Analysis 1: Comparison: Dapagliflozin 10mg/ Dapagliflozin 10mg vs Placebo/ Dapagliflozin 10mg; Test type: Superiority; p = 0.056, Fisher's exact test; Mean Difference (Final Values) = 20.83, 95% CI 2-sided [0.50 to 41.11]

ADVERSE EVENTS:
Time Frame: Up to a maximum of 56 weeks
Arm/Group | Dapagliflozin 10mg/ Dapagliflozin 10mg | Placebo/ Dapagliflozin 10mg
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/33
Serious Adverse Events (participants affected / at risk) | 2/39 | 3/33
Other Adverse Events (participants affected / at risk) | 24/39 | 19/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin 10mg/ Dapagliflozin 10mg (N=39) | Placebo/ Dapagliflozin 10mg (N=33)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin 10mg/ Dapagliflozin 10mg (N=39) | Placebo/ Dapagliflozin 10mg (N=33)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (3)
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (4)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (2)
Fungal infection (Infections and infestations) | 2 (3) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 2 (3)
Pharyngitis streptococcal (Infections and infestations) | 2 (2) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1)
Weight increased (Investigations) | 2 (2) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Vitamin D deficiency (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 5 (6) | 4 (4)
Microalbuminuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT02725593/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT02725593/SAP_001.pdf